CLINICAL TRIAL: NCT04060732
Title: Feasibility and Safety of "Flash Glucose Monitoring-FGM" in an Adult and Selected Pediatric Population.
Brief Title: Feasibility and Safety of "Flash Glucose Monitoring-FGM" in an Adult Italian Population.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Principal Investigator, Riccardo Bonadonna, Director of Endocrinology and Metabolic disease Unit, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 44771
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Flash Glucose Monitoring; Glucose Monitoring; Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Flash Glucose Monitoring Device: The Flash Glucose Monitoring-FGM is a real-time glycemic monitoring system called "hybrid" used by Diabetes Mellitus type 1 patients.
  Interventions: Device: Flash Glucose Monitoring-FGM

INTERVENTIONS:
Device: Flash Glucose Monitoring-FGM — The Flash Glucose Monitoring-FGM is a real-time glycemic monitoring system called "hybrid" will be assigned to the enrolled patients at baseline until the end of follow-up after 12 months.

SUMMARY:
Diabetes is reaching epidemic proportions and a targeted glucose control is key to prevent microvascular complications as well as long-term macrovascular disease.

Self-monitoring of blood glucose (SMBG) in type 1 diabetes (T1D) is mandatory to implement safe and effective adjustments in insulin therapy in order to reduce glucose levels and prevent hypoglycemic episodes. It is known that a higher rate of glucose testing (up to 8 times/day) is associated with improved glucose control, however, long-term repeated daily glucose tests are painful, inconvenient and difficult to pursue.

Continuous glucose monitoring (CGM) is an alternative to SMBG, but the use of conventional CGM has been limited by the need of repeated calibration using capillary glucose testing, relatively short sensor lifespan and high costs. The recently introduced CGM FreeStyle Libre™ (Abbott Diabetes Care, Witney, UK) flash glucose monitoring (FGM), a new generation of glucose testing device, has the advantage to be user friendly by just scanning the reader over the sensor.

The FGM system does not require calibration, has a long sensor lifetime of 14 days and it's relatively affordable, explaining the widespread use of the device.

The Flash Glucose Monitoring-FGM is a real-time glycemic monitoring system called "hybrid" as it is not equipped with alarms capable of alerting the patient to cut-off value for the hypo- or hyperglycemia, but allows the glycemic trend to be viewed at request.

DETAILED DESCRIPTION:
Patients will be identified and enrolled in the Diabetes Departments of different hospitals/clinics in the Emilia Romagna region, Italy. Patients will be divided in two groups A (naive patients,) and B (patients already using the device at enrollment) and followed for 12 months.

Study design is observational prospective and includes 3-months follow up visits until the 12-month final evaluation.

At each visit, patient clinical data, adherence and side effects will be recorded and data download from the device will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes Mellitus type 1 for at least 12 months
* Multi-injection insulin therapy
* C-peptide <0.2 nmol/L
* At least 1 documented episode in the last 12 months of hospitalization (emergency room or ordinary hospitalization) for severe hypoglycemia; hospitalization (emergency room. or ordinary hospitalization) for diabetic ketoacidosis; documented severe hypoglycemia (i.e. with blood glucose measurement).

Exclusion Criteria:

* Diabetes Mellitus type 2
* Other types of diabetes
* Other diseases (excluding endocrinopathies, hypertension and dyslipidemia) that required chronic intake of drugs that may interfere with the glucose-insulin system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of Diabetes Mellitus type 1 for at least 12 months and in multi-injection insulin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Severe hypoglycemia rate | 12 months
  Frequency (number) of serious episodes of hypoglycemia (as defined by the American Diabetes Association, as severe cognitive impairment requiring external assistance for recovery).
Severe hypoglycemia rate | 12 months
  Percentage (%) of patients with at least 1 episode of severe hypoglycemia.

SECONDARY OUTCOMES:
Glucose control | 12 months
  HbA1c (mmol/mol) change from baseline.
Glucose control | 12 months
  Time in hypoglycemia (<3.9 mmol/L) at any time of day.
Glucose control | 12 months
  Time spent with hypoglycemia (<3.1 mmol/L) at any time of day.
Glucose control | 12 months
  Time spent with hypoglycemia (<2.2 mmol/L) at any time of day.
Glucose control | 12 months
  Time spent within the euglycemic range (3.9 - 9.9 mmol/L) at any time of day.
Glucose control | 12 months
  Time spent with hyperglycemia (>10 mmol/L)at any time of day.
Glucose control | 12 months
  Time spent in hyperglycemia (>13.3 mmol/L) at any time of day.
Flash Glucose Monitoring treatment satisfaction | 12 months
  Change in Diabetes Quality Of Life- DQOL score from baseline.
  The original DQOL is a 60-item instrument to assess the diabetes-related QOL of participants. The instrument provides an overall scale score, as well as four subscale scores for 1) satisfaction with treatment, 2) impact of treatment, 3) worry about the future effects of diabetes, and 4) worry about social/vocational issues.
  Items are scored on a 5-point Likert scale and are of two general formats. One format asks about the frequency of negative impact of diabetes itself or of the diabetes treatment and provides response options from 1 (never) to 5 (all the time). The second format asks about satisfaction with treatment and quality of life and is scored from 1 (very satisfied) to 5 (very dissatisfied).
  Higher scores on DQOL items and subscales are, therefore, negatively valenced, indicating problem frequency or dissatisfaction.
Safety of the device | 12 months
  Number (n) of allergic patch reactions.
Feasibility of the device | 12 months
  Number (n) of untimely detachments of the device.
Feasibility of the device | 12 months
  Percentage (%) of recorded data by the device.
Feasibility of the device | 12 months
  Number (n) of device interruptions.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonadonna, MD, Principal Investigator — Regione Emilia-Romagna
Locations (1):
- Azienda Ospedaliero Universitaria, Parma, Italy

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] American Diabetes Association. 6. Glycemic Targets. Diabetes Care. 2017 Jan;40(Suppl 1):S48-S56. doi: 10.2337/dc17-S009. No abstract available. PMID 27979893
- [Background] Miller KM, Beck RW, Bergenstal RM, Goland RS, Haller MJ, McGill JB, Rodriguez H, Simmons JH, Hirsch IB; T1D Exchange Clinic Network. Evidence of a strong association between frequency of self-monitoring of blood glucose and hemoglobin A1c levels in T1D exchange clinic registry participants. Diabetes Care. 2013 Jul;36(7):2009-14. doi: 10.2337/dc12-1770. Epub 2013 Feb 1. PMID 23378621
- [Background] Hoss U, Budiman ES, Liu H, Christiansen MP. Feasibility of Factory Calibration for Subcutaneous Glucose Sensors in Subjects With Diabetes. J Diabetes Sci Technol. 2014 Jan;8(1):89-94. doi: 10.1177/1932296813511747. Epub 2014 Jan 1. PMID 24876543
- [Background] Bailey T, Bode BW, Christiansen MP, Klaff LJ, Alva S. The Performance and Usability of a Factory-Calibrated Flash Glucose Monitoring System. Diabetes Technol Ther. 2015 Nov;17(11):787-94. doi: 10.1089/dia.2014.0378. Epub 2015 Jul 14. PMID 26171659
- [Background] New JP, Ajjan R, Pfeiffer AF, Freckmann G. Continuous glucose monitoring in people with diabetes: the randomized controlled Glucose Level Awareness in Diabetes Study (GLADIS). Diabet Med. 2015 May;32(5):609-17. doi: 10.1111/dme.12713. Epub 2015 Feb 20. PMID 25661981
- [Background] Bonora B, Maran A, Ciciliot S, Avogaro A, Fadini GP. Head-to-head comparison between flash and continuous glucose monitoring systems in outpatients with type 1 diabetes. J Endocrinol Invest. 2016 Dec;39(12):1391-1399. doi: 10.1007/s40618-016-0495-8. Epub 2016 Jun 10. PMID 27287421
- [Derived] Dei Cas A, Aldigeri R, Bellei G, Raffaeli D, Di Bartolo P, Sforza A, Marchesini G, Ciardullo AV, Manicardi V, Bianco M, Monesi M, Vacirca A, Cimicchi MC, Sordillo PA, Altini M, Fantuzzi F, Bonadonna RC; Flash-glucose monitoring Emilia Romagna Regional network. Effectiveness of the flash glucose monitoring system in preventing severe hypoglycemic episodes and in improving glucose metrics and quality of life in subjects with type 1 diabetes at high risk of acute diabetes complications. Acta Diabetol. 2024 Sep;61(9):1177-1184. doi: 10.1007/s00592-024-02298-x. Epub 2024 Jun 4. PMID 38833007